CLINICAL TRIAL: NCT02047630
Title: Efficacy of the Brand-name Latanoprost and One of Its Generic Version in Primary Open Angle Glaucoma and Ocular Hypertension
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Problem with IP supply
Sponsor: CHU de Quebec-Universite Laval (Other)
Responsible Party: Principal Investigator, Marie-Josée Fredette, MD, FRCSC, CHU de Quebec-Universite Laval
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C13-11-1242
Record Dates: First submitted 2014-01-19; First posted 2014-01-28 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Primary Open Angle Glaucoma; Ocular Hypertension
Keywords: Primary open angle glaucoma; Ocular hypertension; latanoprost; generic; intraocular pressure
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Generic latanoprost (Experimental): 1 eye drop hs
  Interventions: Drug: Generic latanoprost; Drug: Brand-name latanoprost
- Brand-name latanoprost (Active Comparator): 1 eye drop hs
  Interventions: Drug: Generic latanoprost; Drug: Brand-name latanoprost

INTERVENTIONS:
Drug: Generic latanoprost
Drug: Brand-name latanoprost
  Other Names: Xalatan

SUMMARY:
The purpose of this study is to evaluate and compare efficacy and tolerability of the brand-name latanoprost and one of its generic version in subjects with primary open angle glaucoma or ocular hypertension.

This randomized, double-blinded, cross-over design study has a 4 months follow-up. There are two periods of 8 weeks. During the first period, subjects put brand-name latanoprost in one eye and the generic version in the other one. In the second period, drops are switched from one eye to the other. There are intraocular pressure measurements (diurnal curves) on day 0 (before treatment), at 8 weeks (at the end of first period) and at 16 weeks (at the end of second period). Variations of intraocular pressure in each eye will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. >18 years old
2. Primary open angle glaucoma, glaucoma suspect or ocular hypertension
3. Bilateral
4. Without any treatment or treated with latanoprost or another prostaglandin analog
5. Intraocular pressure >21mmHg (without treatment or after a washout period)

Exclusion Criteria:

1. Intraocular pressure >30mmHg
2. Secondary glaucoma (uveitic, neovascular, traumatic ) or congenital glaucoma
3. Pseudoexfoliation syndrome
4. Pigmentary dispersion syndrome or Pigmentary glaucoma
5. Severe glaucoma; Cup-to-disc ratio ≥9/10 OU Loss of central visual field (central 10°)
6. Use of other topical medication to lower intraocular pressure
7. Pregnancy and breast-feeding
8. Being allergic to latanoprost or benzalkonium chloride (BAK)
9. Current use of acetazolamide (Diamox)
10. Changes of systemic doses of beta-blockers during study
11. Recent use of topical corticosteroids (<1 month)
12. Contact lens wearer
13. Closed angle at gonioscopy or past angle closure glaucoma
14. Filtration surgery (example. : trabeculectomy)
15. Selective Laser Trabeculoplasty (SLT) or Argon Laser Trabeculoplasty(ALT)
16. Recent Intraocular surgery (<3 months)
17. Refractive surgery
18. Recent iridotomy or capsulotomy (<3 months)
19. Past medical history of ocular trauma (example : angle recession)
20. Past or active uveitis
21. Herpetic keratitis
22. Monocular vision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2014-01; Primary Completion 2014-12-04 (Actual); Study Completion 2014-12-04 (Actual)

PRIMARY OUTCOMES:
Change in Intraocular Pressure (IOP) | 8 weeks, 16 weeks
  Goldman applanation tonometry will be used to measure IOP.

SECONDARY OUTCOMES:
Change in Conjunctival hyperemia | 8 weeks, 16 weeks
Change in corneal staining | 8 weeks, 16 weeks
  Oxford grading scale
Change in TSS-IOP (Treatment Satisfaction Survey for IntraOcular Pressure) | 8 weeks, 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Josée Fredette, MD, FRCSC, Principal Investigator — Centre de recherche du CHU de Québec; Université Laval
Locations (1):
- Centre universitaire d'ophtalmologie, Hôpital du Saint-Sacrement, CHU de Québec, Québec, Canada